CLINICAL TRIAL: NCT01705613
Title: Cost-effectiveness of the Treatment of Attention Deficit/Hyperactivity Disorder With Methylphenidate Immediate-release in Brazil
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, larohde, Luis Augusto Paim Rohde, Hospital de Clinicas de Porto Alegre
Other Study IDs: 100540; 100540 (Other: Comitê de Ética em Pesquisa do Hospital de Clínicas de Porto Alegre (CEP/HCPA)); U1111-1131-1903 (Other: Universal Trial Number)
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Attention Deficit/Hyperactivity Disorder; ADHD; Methylphenidate Immediate-release; Cost-effectiveness; Cost-utility; QALYs
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The first objective is to measure the QALYs (Quality Adjusted Life Years) of Brazilian children and adolescents, submitted to methylphenidate immediate-release treatment for Attention Deficit Hyperactivity Disorder (ADHD). For this, the Health Utility Index scale (HUI) will be completed by the patient and/or family, in two moments of an observation study with immediate-release methylphenidate: at the baseline and 6th month of treatment in the follow-up. The results provides information to calculate the utility measure and determine the QALYs (Quality Adjusted Life Years). After this, for the cost-effectiveness of the treatment, it will be used a Markov model of decision analysis, and a Monte Carlo simulation with 10,000 random trials.

Subjects will be submitted to immediate-release methylphenidate treatment in a maximum dose of 0.5mg/kg/day. The total treatment monitoring is 06 (six) months, and patients will be evaluated at baseline, first, third and sixth month. The HUI rating scales are fulfilled by parents and patients (if >12 years old only) at baseline and 6th month. The period for inclusion of new patients comprises from 01/01/2011 to 31/12/2013.

DETAILED DESCRIPTION:
Currently, Brazil has no estimates for quality of life, and/or utilities for ADHD economy analysis. Such data is necessary to calculate the QALYs (Quality Adjusted Life Years). Thus, the investigators will implement the Health Utility Index tool (HUI) to be completed by the patient and/or family, in two moments of an observational study with immediate-release methylphenidate: at baseline and 6th month of treatment. The determination of the QALY as an outcome in the decision analysis is justified because HUI incorporates into a single measure morbidity and mortality. The results of the cost-effectiveness study will assist government agencies in the process of decision making.

To determine the cost-effectiveness of methylphenidate immediate release available in the Brazilian market, the investigators will use a Markov model of decision analysis. The development of the model and analysis of the results will adopt the standards established in the Methodological Guidelines of the Brazilian Ministry of Health, and the perspective will be of the Brazilian National Health System. Medications prices will be obtained through the Board of Market Regulation of Medicines (CMED) at the site of ANVISA (National Health Surveillance Agency). For the treatment strategy that provides greatest cost ratio it will be calculated the incremental cost-effectiveness, compared to the lower cost. To estimate more accurately the impact on life, a Monte Carlo simulation with 10,000 random trials will be conducted.

This is a one treatment group and observational study, with 140 patients, and no controls. Where indicated, it will be suggested the use of 10 mg methylphenidate in a maximum dose of 0.5 mg / kg / day. The total treatment monitoring is 06 (six) months, and patients will be evaluated at baseline, first, third and sixth month. The HUI rating scales will be fulfilled by parents and patients (if >12 years old only) at baseline and 6th month. The period for inclusion of new patients comprises from 01/01/2011 to 31/12/2013.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of attention deficit/hyperactivity disorder with impairment
* Children and adolescents (age from 06 to 18 years old)
* absence of contraindication for the use of methylphenidate immediate release

Exclusion Criteria:

* Contraindication methylphenidate immediate release use
* Neurological diseases
* Discordance with the informed consent form
* IQ<70
* Neurological diseases

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with indication of Attention Deficit/Hyperactivity Disorder treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Swanson, Nolan, and Pelham Rating Scale (SNAP-IV) | Baseline, 1th, 3rd and 6th month
Health Utility Index | Baseline and 6th month

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Rohde, MD, PhD, Study Chair — Hospital de Clinicas de Porto Alegre; Carlos R Moreira Maia, MD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Maia CR, Stella SF, Wagner F, Pianca TG, Krieger FV, Cruz LN, Polanczyk GV, Rohde LA, Polanczyk CA. Cost-utility analysis of methylphenidate treatment for children and adolescents with ADHD in Brazil. Braz J Psychiatry. 2016 Mar;38(1):30-8. doi: 10.1590/1516-4446-2014-1516. Epub 2015 Sep 8. PMID 26375808